CLINICAL TRIAL: NCT00410943
Title: A Randomized, Double-Blind, Repeated Dose, Parallel-Group Comparison of the Efficacy & Tolerability of Dilaudid SR Tablets and Immediate Release Dilaudid Tablets (Hydromorphone HCI) in Patients With Chronic Pain
Brief Title: Study of the Effectiveness and Tolerability of OROS Hydromorphone HCI SR(Slow-release) Tablets and Immediate-Release Hydromorphone Tablets in Patients With Chronic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR013276
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Pain
Keywords: Cancer pain; Oral analgesic; OROS hydromorphone HCI
MeSH Terms: conditions — Pain; Cancer Pain

INTERVENTIONS:
Drug: OROS Hydromorphone HCI SR (slow release)

SUMMARY:
The purpose of this study was to characterize a safe and effective means of conversion and titration to an appropriate dose of hydromorphone HCI, to demonstrate comparable efficacy of OROS hydromorphone HCI SR (slow release) and hydromorphone HCI IR (immediate release) following administration of approximately equivalent total daily doses and demonstrate a significant dose-response relationship between OROS hydromorphone HCI SR (slow release) for breakthrough pain medication use or alternatively, diary-based analgesic scores

DETAILED DESCRIPTION:
This was a randomized (patients are assigned different treatments based on chance), double-blind (neither the patient nor the physician knows whether drug or placebo is being taken, or at what dosage), repeated-dose, three-arm parallel group study conducted in three phases. Following a Prior Opioid Stabilization Phase, wherein patients were required to be on a stable dose of chronic opioid therapy, patients were converted, titrated and stabilized on hydromorphone HCI IR (immediate release) to achieve acceptable levels of analgesia in the Open-Label Hydromorphone HCI IR (immediate release) Conversion, Titration, and Stabilization Phase. Supplementary hydromorphone HCI IR (immediate release) was provided for breakthrough pain, and patients were considered stabilized on hydromorphone HCI IR (immediate release) when the total daily dose of hydromorphone HCI IR (immediate release) remained unchanged with no more than three hydromorphone HCI IR (immediate release) breakthrough pain medication doses per day for 2 consecutive days. Patients who were able to achieve a stable total daily dose of at least 20 mg but not more than 60 mg of hydromorphone HCI IR (immediate release) (exclusive of breakthrough pain medication) within the 14 day Open-Label hydromorphone HCI IR (immediate release) Conversion, Titration, and Stabilization Phase of the study entered the Double-Blind, Randomized, Repeat Dosing Phase of the study. Patients were randomized to receive 7 days of either OROS hydromorphone HCI SR (slow release) at a daily dose approximately equal to their stabilized total daily dose of hydromorphone HCI IR (immediate release), OROS hydromorphone HCI SR (slow release) at a daily dose approximately equal to one-half their stabilized total daily dose of hydromorphone HCI IR (immediate release) (1/2 OROS hydromorphone slow release), or hydromorphone HCI IR (immediate release) at the same daily dose on which they were stabilized (hydromorphone immediate release). Patients who completed the study were eligible for participation in an open-label OROS hydromorphone SR (slow release) long-term extension study (Protocol DO-109). OROS hydromorphone slow release 8, 16 and 32 mg tablets, hydromorphone immediate release 2 and 4 mg tablets, placebo immediate release 2 and 4 mg tablets and placebo slow release 8, 16, and 32 mg tablets taken orally for 7 days

ELIGIBILITY:
Inclusion Criteria:

* Patients who have chronic non-malignant or cancer pain currently receiving strong or transdermal opioid analgesics on a daily basis or patients suitable for advancement of therapy to step 3 on the WHO (World Health Organization) analgesic ladder
* Patients who, at Visit 2, require the equivalent of at least 80 mg but no more than 300 mg of oral morphine sulfate (exclusive of breakthrough pain medication) every 24 hours or at least 25 micrograms an hour but no more than 75 micrograms an hour of Fentanyl
* Patients must be on a stable dose of a strong opioid medication at Visit 2. Patients will be considered stabilized when the total daily dose of their prestudy opioid medication remains unchanged, with no more than three opioid breakthrough pain doses/day administered for breakthrough pain, for two consecutive days
* Patients who can be expected to have reasonably stable opioid requirements for the duration of the study

Exclusion Criteria:

* Patients intolerant of or hypersensitive to hydromorphone (or other opioid agonists)
* Patients who have difficulty swallowing or are unable to swallow tablets
* Patients who are pregnant or breast-feeding. Female patients of child-bearing potential must be following a medically recognized contraceptive program prior to and during the study. A negative pregnancy test is required prior to administration of study drug
* Patients with any gastrointestinal disorder, including pre-existing severe gastrointestinal narrowing that may affect the absorption or transit of orally administered drugs
* Patients with any intracranial lesion, increased intracranial pressure, seizure disorder, stroke within the past 6 months, and disorders of cognition
* Patients with clinically significant impaired kidney or liver function, thyroid disease, enlarged prostate, or urethral narrowing
* Patients who may be at risk for serious decreases in blood pressure upon administration of an opioid analgesic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Study Completion 1999-06 (Actual)

PRIMARY OUTCOMES:
This study demonstrated a dose-response relationship with OROS hydromorphone slow release and no statistically significant differences in efficacy results between OROS hydromorphone slow release and immediate release at approximately equal doses.

SECONDARY OUTCOMES:
There were no statistically significant differences between treatment groups in measures of efficacy at baseline or endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA